CLINICAL TRIAL: NCT05223777
Title: KINCISE™ Surgical Automated System in Total Hip Arthroplasty (THA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Todd Kelley, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS20004 IRB 2020-0656
Record Dates: First submitted 2021-07-01; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Osteoarthritis, Hip
Keywords: total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Patients will undergo primary total hip athroplasties through a direct anterior surgical approach using press fit implants. Anesthesia will be either general anesthesia or spinal anesthesia.Multimodal analgesia and rapid recovery techniques are used for all procedures. Twenty-five (25) of these procedures will be performed using the KINCISE and 25 will be performed using traditional handheld mallets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- KINCISE (Active Comparator): The KINCISE™ Surgical Automated System (KINCISE) (DePuy Synthes Products, Inc, Warsaw, IN) was developed to replace the handheld mallet traditionally used in total hip arthroplasty (THA). The device is an FDA-approved medical instrument. As such, the focus of the study does not relate to the safety and efficacy of the device, which has already been established. Instead, the current IRB proposal investigates whether there are long-term benefits to patient outcomes that differ between KINCISE-guided versus mallet THA.
  Interventions: Device: KINCISE
- Traditional Mallet (Placebo Comparator): A traditional mallet will be used during surgery in this group.
  Interventions: Device: Traditional Handheld Mallet

INTERVENTIONS:
Device: KINCISE — The KINCISE™ Surgical Automated System (KINCISE) (DePuy Synthes Products, Inc, Warsaw, IN) was developed to replace the handheld mallet traditionally used in total hip arthroplasty (THA). The device is an FDA-approved medical instrument.
  Arms: KINCISE
Device: Traditional Handheld Mallet — The handheld mallet traditionally used in total hip arthroplasty.
  Arms: Traditional Mallet

SUMMARY:
There is a growing interest in the effects of mental health and wellness on orthopedic intervention outcomes, not only in terms of how advances in surgical procedures influence patient outcomes, but also with regard for physician physical and mental well-being. Although total hip arthroplasty (THA) is associated with favorable clinical outcomes as assessed by surgeon evaluation, radiographic analysis and implant longevity, unfavorable long-term pain and quality of life outcomes are consistently observed in upwards of 20% of patients receiving THAs. As such, the need to understand and address the determinants of positive and negative outcomes is of critical importance if the field hopes to continue to advance strategies to improve long-term outcomes for joint replacement. The overarching goal of this application is to assess the benefits of the KINCISE for patient recovery outcomes related to physical and mental well-being.

DETAILED DESCRIPTION:
Participants. Participants (N= 50) will be recruited from the Department of Orthopaedic Surgery service at the University of Cincinnati Medical Center. The service refers approximately 240 patients for conventional THA annually, approximately 190 of which are performed by the PI. All participants will be paid for their participation.

Clinical and Behavioral Assessments. Throughout the proposed work, we intend to examine patient recovery time, long-term pain outcomes, mood, and sleep habits. Assessments for pain, functionality, anxiety, and depression, will be administered electronically to each patient at study onset and conclusion using standardized psychological scales. Completion time for these psychological assessments is approximately 30 minutes.

Phase 1: Preoperative Assessment (6 weeks prior to day of surgery). All patients will complete a study entrance exam consisting of clinical assessments of joint and pain functionality (HSS) and behavioral assessments of patient-reported general health (SF-36), joint pain and functionality (HOOS), anxiety (GAD-7), and depression (PHQ-9). Completion time for these assessments is approximately 30 minutes. Participants will also have the passive, automatic sensing app (Mae) installed on their smartphone to measure sleep habits, physical activity, social interaction, and mood. The app will collect passive sensing data and deliver the 3-minute weekly survey (as described above) throughout the entirety of the study.

Phase 2: Surgical Intervention. Patients will undergo primary THAs through a direct anterior surgical approach using press fit implants. Anesthesia will be either general anesthesia or spinal anesthesia. Multimodal analgesia and rapid recovery techniques are used for all procedures. Twenty-five (25) of these procedures will be performed using the KINCISE and 25 will be performed using traditional handheld mallets. Patients will be pseudorandomly assigned to KINCISE or handheld mallet conditions to match for patient age, sex, and preoperative functionality and pain scores. Assignments to treatment conditions will be counterbalanced to account for the number of TJAs performed each day by the surgeon. All surgeries will be recorded using a high definition digital camera compatible for use in OS#, UC IRB 2020-XXXXVersion 1.0 pg. 5 surgical suites. The camera will be positioned so as not to record the patient's face. Video and audio recording will be used to calculate broach time, total length of each procedure, and mallet strikes.

Phase 3: Postoperative Longitudinal Study of Sleep, Mood, and Pain. Patients will be followed longitudinally for one year after surgery. During this phase, sleep habits, physical activity, social interaction, and mood data will continue to be collected and weekly assessments of mood, functionality, and pain will continue to be administered using the Mae smartphone app. Post-operative clinical assessments (HHS) and patient reports of joint pain and functionality (HOOS) will be administered and collected at six weeks, three months, and one year for all patients. At the one-year time point, patients will additionally complete full versions of the SF-36, the PHQ-9 depression scale, and the GAD-7 anxiety scale. Of interest is whether KINCISE-guided procedures result in more favorable recovery times and pain outcomes and whether such changes are accompanied by improved sleep quality and reduced anxiety and depression. Because Mae employs continuous data collection through passive sensing and weekly surveys, the research project offers a unique opportunity to study the duration of improvements in functionality and pain reduction at a level of granularity that cannot be accomplished by periodic office follow-ups alone (e.g., when do patients reach/surpass their preoperative walking speed?).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants over age 21 with a compatible smartphone (Apple iPhone 6s or newer running iOS 13 or higher) are eligible to participate.
* Participants must be community ambulatory

Exclusion Criteria:

* Age less than 21.
* Incompatible smartphone device.
* History of neurological injury or pathology.
* Prior total joint athroplasty in the preceding year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The Short Form (36) Health Survey | 1 year
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

SECONDARY OUTCOMES:
The Patient Health Questionnaire20 (PHQ-9) | 1 year
  Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Kelley, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Univrsity of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKinney RE Jr. The Daunting Career of the Physician-Investigator. Acad Med. 2017 Oct;92(10):1368-1370. doi: 10.1097/ACM.0000000000001869. PMID 28767494
- [Background] Erickson SM, Rockwern B, Koltov M, McLean RM; Medical Practice and Quality Committee of the American College of Physicians. Putting Patients First by Reducing Administrative Tasks in Health Care: A Position Paper of the American College of Physicians. Ann Intern Med. 2017 May 2;166(9):659-661. doi: 10.7326/M16-2697. Epub 2017 Mar 28. PMID 28346948
- [Background] Shanafelt TD, Dyrbye LN, Sinsky C, Hasan O, Satele D, Sloan J, West CP. Relationship Between Clerical Burden and Characteristics of the Electronic Environment With Physician Burnout and Professional Satisfaction. Mayo Clin Proc. 2016 Jul;91(7):836-48. doi: 10.1016/j.mayocp.2016.05.007. Epub 2016 Jun 27. PMID 27313121
- [Background] Kuhn T, Basch P, Barr M, Yackel T; Medical Informatics Committee of the American College of Physicians. Clinical documentation in the 21st century: executive summary of a policy position paper from the American College of Physicians. Ann Intern Med. 2015 Feb 17;162(4):301-3. doi: 10.7326/M14-2128. PMID 25581028
- [Background] Babbott S, Manwell LB, Brown R, Montague E, Williams E, Schwartz M, Hess E, Linzer M. Electronic medical records and physician stress in primary care: results from the MEMO Study. J Am Med Inform Assoc. 2014 Feb;21(e1):e100-6. doi: 10.1136/amiajnl-2013-001875. Epub 2013 Sep 4. PMID 24005796
- [Background] Kelley TC, Adams MJ, Mulliken BD, Dalury DF. Efficacy of multimodal perioperative analgesia protocol with periarticular medication injection in total knee arthroplasty: a randomized, double-blinded study. J Arthroplasty. 2013 Sep;28(8):1274-7. doi: 10.1016/j.arth.2013.03.008. Epub 2013 Apr 20. PMID 23608085
- [Background] Kelley TC, Tucker KK, Adams MJ, Dalury DF. Use of tranexamic acid results in decreased blood loss and decreased transfusions in patients undergoing staged bilateral total knee arthroplasty. Transfusion. 2014 Jan;54(1):26-30. doi: 10.1111/trf.12167. Epub 2013 Mar 22. PMID 23521109
- [Background] Dalury DF, Kelley TC, Adams MJ. Modern proximally tapered uncemented stems can be safely used in Dorr type C femoral bone. J Arthroplasty. 2012 Jun;27(6):1014-8. doi: 10.1016/j.arth.2011.12.019. Epub 2012 Feb 8. PMID 22325961
- [Background] Dalury DF, Tucker KK, Kelley TC. All-polyethylene tibial components in obese patients are associated with low failure at midterm followup. Clin Orthop Relat Res. 2012 Jan;470(1):117-24. doi: 10.1007/s11999-011-1964-1. PMID 21739322
- [Background] Dalury DF, Tucker KK, Kelley TC. When can I drive?: brake response times after contemporary total knee arthroplasty. Clin Orthop Relat Res. 2011 Jan;469(1):82-6. doi: 10.1007/s11999-010-1507-1. PMID 20700671
- [Background] Huckins JF, daSilva AW, Wang R, Wang W, Hedlund EL, Murphy EI, Lopez RB, Rogers C, Holtzheimer PE, Kelley WM, Heatherton TF, Wagner DD, Haxby JV, Campbell AT. Fusing Mobile Phone Sensing and Brain Imaging to Assess Depression in College Students. Front Neurosci. 2019 Mar 21;13:248. doi: 10.3389/fnins.2019.00248. eCollection 2019. PMID 30949024
- [Background] Koutsouleris N, Dwyer DB, Degenhardt F, Maj C, Urquijo-Castro MF, Sanfelici R, Popovic D, Oeztuerk O, Haas SS, Weiske J, Ruef A, Kambeitz-Ilankovic L, Antonucci LA, Neufang S, Schmidt-Kraepelin C, Ruhrmann S, Penzel N, Kambeitz J, Haidl TK, Rosen M, Chisholm K, Riecher-Rossler A, Egloff L, Schmidt A, Andreou C, Hietala J, Schirmer T, Romer G, Walger P, Franscini M, Traber-Walker N, Schimmelmann BG, Fluckiger R, Michel C, Rossler W, Borisov O, Krawitz PM, Heekeren K, Buechler R, Pantelis C, Falkai P, Salokangas RKR, Lencer R, Bertolino A, Borgwardt S, Noethen M, Brambilla P, Wood SJ, Upthegrove R, Schultze-Lutter F, Theodoridou A, Meisenzahl E; PRONIA Consortium. Multimodal Machine Learning Workflows for Prediction of Psychosis in Patients With Clinical High-Risk Syndromes and Recent-Onset Depression. JAMA Psychiatry. 2021 Feb 1;78(2):195-209. doi: 10.1001/jamapsychiatry.2020.3604. PMID 33263726
- [Background] Neta M, Norris CJ, Whalen PJ. Corrugator muscle responses are associated with individual differences in positivity-negativity bias. Emotion. 2009 Oct;9(5):640-8. doi: 10.1037/a0016819. PMID 19803586
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. CMAJ. 2012 Feb 21;184(3):E191-6. doi: 10.1503/cmaj.110829. Epub 2011 Dec 19. PMID 22184363
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Lowe B, Wahl I, Rose M, Spitzer C, Glaesmer H, Wingenfeld K, Schneider A, Brahler E. A 4-item measure of depression and anxiety: validation and standardization of the Patient Health Questionnaire-4 (PHQ-4) in the general population. J Affect Disord. 2010 Apr;122(1-2):86-95. doi: 10.1016/j.jad.2009.06.019. Epub 2009 Jul 17. PMID 19616305
- [Background] Lemke MR, Wendorff T, Mieth B, Buhl K, Linnemann M. Spatiotemporal gait patterns during over ground locomotion in major depression compared with healthy controls. J Psychiatr Res. 2000 Jul-Oct;34(4-5):277-83. doi: 10.1016/s0022-3956(00)00017-0. PMID 11104839
- [Background] Kriegeskorte N, Mur M, Bandettini P. Representational similarity analysis - connecting the branches of systems neuroscience. Front Syst Neurosci. 2008 Nov 24;2:4. doi: 10.3389/neuro.06.004.2008. eCollection 2008. PMID 19104670